CLINICAL TRIAL: NCT00397358
Title: Open-label Study to Evaluate the Effects of Once Daily Extraneal (7.5% Icodextrin) Peritoneal Dialysis Solution on Triglyceride Levels in Peritoneal Dialysis Patients
Brief Title: Effect of Extraneal (Icodextrin)on Triglyceride Levels in PD Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31656
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Peritoneal Dialysis; Hypertriglyceridemia
Keywords: Peritoneal Dialysis; Hypertriglyceridemia; Extraneal(7.5% icodextrin)Peritoneal Dialysis Solution
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Icodextrin; Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Extraneal (7.5% icodextrin) Peritoneal Dialysis Solution

SUMMARY:
This is a Phase IV study evaluating triglyceride levels in peritoneal dialysis patients.

DETAILED DESCRIPTION:
This prospective, open label, multi-center study evaluates the use of 7.5% icodextrin used in the long-dwell exchange in peritoneal dialysis patients with elevated triglyceride levels. Fasting triglyceride levels will be measured during the study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* CAPD/APD on dialysis for at least 3 months
* Elevated fasting triglyceride levels

Exclusion Criteria:

* enrolled in another study requiring IRB approval
* allergy to starch-based polymers
* glycogen storage disease
* maltose or isomaltose intolerance
* active alcohol/substance abuse
* Pregnant or nursing
* received an investigational drug within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting triglyceride levels.

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Healthcare Corporation, Study Director — Call central contact for information
Locations (3):
- United States (3):
  - Kaiser Santa Clara - Homestead, Santa Clara, California
  - Nephrology Specialists, Michigan City, Indiana
  - Dialysis Center of Lincoln, Lincoln, Nebraska

REFERENCES:
- [Background] Holmes CJ, Shockley TR. Strategies to reduce glucose exposure in peritoneal dialysis patients. Perit Dial Int. 2000;20 Suppl 2:S37-41. PMID 10911641
- [Background] Bredie SJ, Bosch FH, Demacker PN, Stalenhoef AF, van Leusen R. Effects of peritoneal dialysis with an overnight icodextrin dwell on parameters of glucose and lipid metabolism. Perit Dial Int. 2001 May-Jun;21(3):275-81. PMID 11475343
- [Background] Martikainen T, Teppo AM, Gronhagen-Riska C, Ekstrand A. Benefit of glucose-free dialysis solutions on glucose and lipid metabolism in peritoneal dialysis patients. Blood Purif. 2005;23(4):303-10. doi: 10.1159/000086553. Epub 2005 Jun 23. PMID 15980620
- [Background] Kronenberg F, Lingenhel A, Neyer U, Lhotta K, Konig P, Auinger M, Wiesholzer M, Andersson H, Dieplinger H. Prevalence of dyslipidemic risk factors in hemodialysis and CAPD patients. Kidney Int Suppl. 2003 May;(84):S113-6. doi: 10.1046/j.1523-1755.63.s84.23.x. PMID 12694323
- [Background] Amici G, Orrasch M, Da Rin G, Bocci C. Hyperinsulinism reduction associated with icodextrin treatment in continuous ambulatory peritoneal dialysis patients. Adv Perit Dial. 2001;17:80-3. PMID 11510303
- [Background] Furuya R, Odamaki M, Kumagai H, Hishida A. Beneficial effects of icodextrin on plasma level of adipocytokines in peritoneal dialysis patients. Nephrol Dial Transplant. 2006 Feb;21(2):494-8. doi: 10.1093/ndt/gfi197. Epub 2005 Oct 12. PMID 16221697